CLINICAL TRIAL: NCT00016380
Title: A Randomized Phase III Double-Blind Study Of Ondansetron And Dexamethasone Versus Ondansetron And Placebo In The Prophylaxis Of Radiation-Induced Emesis
Brief Title: Ondansetron With/Out Dexamethasone to Prevent Vomiting in Patients Receiving Radiation to the Upper Abdomen
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: NCIC Clinical Trials Group (Network)
Responsible Party: Sponsor
Organization: Canadian Cancer Trials Group (Network)
Allocation: Randomized | Masking: None | Purpose: Supportive Care
Other Study IDs: SC19; CAN-NCIC-SC19 (Other: PDQ); CDR0000068627 (Other: PDQ)
Record Dates: First submitted 2001-05-06; First posted 2003-01-27 (Estimated); Last update posted 2020-04-03 (Actual); Status verified 2020-04

CONDITIONS: Cancer
Keywords: nausea and vomiting; stage I colon cancer; stage II colon cancer; stage III colon cancer; stage IV colon cancer; stage I gastric cancer; stage II gastric cancer; stage III gastric cancer; stage IV gastric cancer; recurrent gastric cancer; stage I pancreatic cancer; stage II pancreatic cancer; stage III pancreatic cancer; recurrent pancreatic cancer; recurrent colon cancer; recurrent cervical cancer; stage IB cervical cancer; stage IIB cervical cancer; stage IVB cervical cancer; stage IA cervical cancer; stage IIA cervical cancer; stage IVA cervical cancer; stage I ovarian epithelial cancer; stage II ovarian epithelial cancer; stage III ovarian epithelial cancer; stage IV ovarian epithelial cancer; recurrent ovarian epithelial cancer; localized gastrointestinal carcinoid tumor; regional gastrointestinal carcinoid tumor; metastatic gastrointestinal carcinoid tumor; recurrent gastrointestinal carcinoid tumor; localized resectable adult primary liver cancer; localized unresectable adult primary liver cancer; advanced adult primary liver cancer; recurrent adult primary liver cancer; small intestine adenocarcinoma; small intestine lymphoma; small intestine leiomyosarcoma; localized gallbladder cancer; unresectable gallbladder cancer; recurrent gallbladder cancer; localized extrahepatic bile duct cancer; unresectable extrahepatic bile duct cancer; recurrent extrahepatic bile duct cancer; recurrent small intestine cancer; testicular seminoma; carcinoma of the appendix; quality of life; stage IV pancreatic cancer
MeSH Terms: conditions — Neoplasms; Nausea; Vomiting; Colonic Neoplasms; Stomach Neoplasms; Pancreatic Neoplasms; Uterine Cervical Neoplasms; Carcinoma, Ovarian Epithelial; Carcinoma, Hepatocellular; Gallbladder Neoplasms; Bile Duct Neoplasms; Seminoma; Appendiceal Neoplasms | interventions — Dexamethasone; Ondansetron

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: dexamethasone
Drug: ondansetron
Procedure: quality-of-life assessment

SUMMARY:
RATIONALE: Antiemetic drugs may help to reduce or prevent vomiting in patients treated with radiation therapy. It is not yet known if ondansetron is more effective with or without dexamethasone in preventing vomiting caused by radiation therapy.

PURPOSE: This randomized phase III trial is comparing how well ondansetron works with or without dexamethasone in preventing vomiting in patients with cancer who are receiving radiation therapy to the upper abdomen.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the effectiveness of ondansetron with or without dexamethasone as prophylaxis for radiation-induced emesis and nausea in patients receiving upper abdominal radiotherapy.
* Compare toxicity of these regimens in these patients.
* Compare quality of life of patients treated with these regimens.

OUTLINE: This is a randomized, double-blind, placebo-controlled, multicenter study. Patients are stratified according to radiotherapy field description (whole abdomen and pelvis vs partial abdomen and pelvis vs partial abdomen only). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive oral ondansetron twice daily and oral dexamethasone daily for 5-7 days concurrently with the first 5 fractions of radiotherapy.
* Arm II: Patients receive oral ondansetron twice daily and oral placebo daily for 5-7 days concurrently with the first 5 fractions of radiotherapy.

Treatment continues in both arms in the absence of disease progression or unacceptable toxicity.

Quality of life is assessed at baseline, prior to starting radiotherapy if more than 5 days since randomization, prior to the 5th and 15th fractions of radiotherapy, and 1 month after completion of radiotherapy.

Patients are followed at 1 month.

PROJECTED ACCRUAL: A total of 100-200 patients (50-100 per arm) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Cancer patients who are scheduled to receive radiotherapy within the next 3 weeks

  * Total dose at least 2,000 cGy delivered in at least 15 fractions
  * 1 fraction per day, 5 days per week
  * Treatment field to include an area of at least 80 cm2 in the anterior/posterior direction encompassing the upper abdomen
* At risk of developing radiation-induced emesis
* No emesis (retching and/or vomiting) or nausea with severity greater than 2 within the past week

PATIENT CHARACTERISTICS:

Age:

* 16 and over

Performance status:

* ECOG 0-3

Life expectancy:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* No jaundice
* No moderate to severe hepatic dysfunction

Renal:

* Not specified

Gastrointestinal:

* No active peptic ulcer
* No lactose intolerance

Other:

* No concurrent condition or illness that contraindicates corticosteroids, serotonin antagonists, or prochlorperazine (e.g., diabetes mellitus)
* No prior unusual or allergic reaction to a serotonin antagonist (ondansetron, dolasetron, or granisetron), corticosteroid, or prochlorperazine
* No condition that would preclude accessibility to treatment or follow-up
* Able and willing to complete diary and quality of life questionnaires in either English or French
* Able to swallow

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* At least 1 week since prior cytotoxic therapy
* No concurrent cytotoxic therapy

Endocrine therapy:

* No concurrent corticosteroids other than topical or inhaled preparations

Radiotherapy:

* See Disease Characteristics
* At least 1 week since prior radiotherapy
* No concurrent cranial radiotherapy

Surgery:

* Not specified

Other:

* At least 2 days since prior medication with antiemetic intent

Ages: 16 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 211 (Actual)
Dates: Start 2001-02-28 (Actual); Primary Completion 2004-04-30 (Actual); Study Completion 2009-02-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Wong, MD, Study Chair — Princess Margaret Hospital, Canada
Locations (14):
- Canada (14):
  - Cross Cancer Institute, Edmonton, Alberta
  - British Columbia Cancer Agency - Centre for the Southern Interior, Kelowna, British Columbia
  - Fraser Valley Cancer Centre at British Columbia Cancer Agency, Surrey, British Columbia
  - British Columbia Cancer Agency, Vancouver, British Columbia
  - Nova Scotia Cancer Centre, Halifax, Nova Scotia
  - Cancer Care Ontario-London Regional Cancer Centre, London, Ontario
  - Northwestern Ontario Regional Cancer Care, Thunder Bay, Ontario
  - Toronto Sunnybrook Regional Cancer Centre, Toronto, Ontario
  - Princess Margaret Hospital, Toronto, Ontario
  - CHUS-Hopital Fleurimont, Fleurimont, Quebec
  - Maisonneuve-Rosemont Hospital, Montreal, Quebec
  - McGill University, Montreal, Quebec
  - Centre Hospitalier de l'Universite de Montreal, Montreal, Quebec
  - Centre Hospitalier Universitaire de Quebec, Québec, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] National Cancer Institute of Canada Clinical Trials Group (SC19); Wong RK, Paul N, Ding K, Whitehead M, Brundage M, Fyles A, Wilke D, Nabid A, Fortin A, Wilson D, McKenzie M, Ackerman I, Souhami L, Chabot P, Pater J. 5-hydroxytryptamine-3 receptor antagonist with or without short-course dexamethasone in the prophylaxis of radiation induced emesis: a placebo-controlled randomized trial of the National Cancer Institute of Canada Clinical Trials Group (SC19). J Clin Oncol. 2006 Jul 20;24(21):3458-64. doi: 10.1200/JCO.2005.04.4685. PMID 16849762
- [Result] Paul N, Wong R, Brundage Michael, et al.: Symptom assessment in SC19: ondansetron plus dexamethasone as prophylaxis against radiation-induced emesis - a National Cancer Institute of Canada Clinical Trials Group (NCIC CTG) study. [Abstract] Support Care Cancer 13 (6): A-04-033, 419, 2005.
- [Result] Paul N, Wong R, Whitehead M, et al.: Daily diary reporting of symptoms in SC19: a National Cancer Institute of Canada Clinical Trials Group (NCIC CTG) study of prophylaxis against radiation-induced emesis. [Abstract] Support Care Cancer 13 (6): A-04-034, 419, 2005.
- [Result] Wong R, Paul N, Ding K, et al.: Optimizing prophylaxis of radiation induced emesis (RIE): a phase III double blind randomized study comparing ondansetron plus dexamethasone (OndDex) vs ondansetron alone (OndPlac). [Abstract] Support Care Cancer 13 (6): A-04-043, 423, 2005.